CLINICAL TRIAL: NCT06405919
Title: Risk of Malignancy in Endemic Long Standing Nodular Goitres: a Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Khartoum (Other)
Collaborators: Sudan Medical Specialization Board (Other Government)
Responsible Party: Principal Investigator, Seifeldin Mahdi, Associate professor of surgery, University of Khartoum
Other Study IDs: UofK
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Incidence of Thyroid Cancer in Long Standing MNG
Keywords: : goitre, long standing, malignant risk, incidental.
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Resected goitres for histopathology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with goitres 10 years or more: Patients with long standing multinodular goitres of 10years or more presenting to surgical unit in Khartoum Teaching Hospital -Sudan. Checking incidence of malignancy in this group.
  Interventions: Diagnostic Test: Histopathology

INTERVENTIONS:
Diagnostic Test: Histopathology — Thyroidectomy for patients and histological examination of specimen to determine incidence of malignancy.

SUMMARY:
To determine the incidence of thyroid cancer in patients with long standing goitres presenting for surgery.

DETAILED DESCRIPTION:
This is a prospective cohort study The objective is to determine the incidence of cancer in patients with long standing goitres( more than 10 years ) who present for surgery in Khartoum Teaching Hopspital - Sudan.

Introduction: goitre is endemic in Sudan with prevalence ranging between 5-42% in different regions of the country. Patients are referred for surgery only if they develop pressure symptoms.

The incidence of thyroid carcinoma is high in endemic goitrous areas. Determining the risk of cancer in patient with long standing goitres may help in early early referral and early surgical intervention.

Methods: This is prospective cohort study including 160 patients with long standing goitrers of 10 years or more who presented from March 2017 to September 2017 to Khartoum Teaching Hospital-Sudan

ELIGIBILITY:
Inclusion Criteria:

* All patients with long standing goitres of 10 years or more

Exclusion Criteria:

* Non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with long standing goitres presenting for surgery in Khartoum Teaching Hospital March 2017-September 2018
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of malignancy | March 2017-September 2018
  Rate of malignancy in resected goitre specimens

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elmakki Abdella, MS,FRCSI, Study Director — University of Khartoum -Faculty of Medicine
Locations (1):
- Faculty of Medicine University of Khartoum, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided